CLINICAL TRIAL: NCT03072680
Title: Efficacy of a Positive Psychology Intervention Through a Mobile App: a Randomized Controlled Trial
Brief Title: Efficacy of a Positive Psychology Intervention Through a Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: University of Twente (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16337
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Not Flourishing Population
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BPS PAST + BPS FUT (Experimental): Participants practice BPS PAST the first week, then they switch fot BPS FUT.
  Interventions: Behavioral: BPS PAST; Behavioral: BPS FUT
- BPS FUT (Experimental): Participants practice BPS FUT during the two weeks.
  Interventions: Behavioral: BPS FUT
- CONTROL (Active Comparator): Participants practice DAILY ACTIVITIES for the two weeks.
  Interventions: Behavioral: DAILY ACTIVITIES

INTERVENTIONS:
Behavioral: BPS PAST — Participants think about themselves in a past when they displayed their best self. Then, they visualize this with the help of audio instructions.
  They will practice within a mobile app.
  Arms: BPS PAST + BPS FUT
Behavioral: BPS FUT — Participants think about themselves in the future after everything has gone as well as it possibly could. Then, they visualize this with the help of audio instructions.
  They will practice within a mobile app.
  Arms: BPS FUT; BPS PAST + BPS FUT
Behavioral: DAILY ACTIVITIES — Participants think about the activities they did during the last 24 hours. Then, they visualize this with the help of audio instructions.
  They will practice within a mobile app.
  Arms: CONTROL

SUMMARY:
The aim of this study is to analyze the efficacy of several variations of an already validated Positive Psychology Intervention (PPI) called Best Possible Self in not flourishing population. This will be done through a mobile app specially designed for this aim.

Concretely, the design will permit to compare the classic intervention (BPS Future), a new variation (BPS Past), and a combination of both components (BPS Past+Future).

Participants will be randomly assigned to one of 3 conditions, in which they will practice the intervention for two weeks:

* BPS-PAST + BPS FUT condition: Participants will practice BPS Past for one week, and then they will switch to BPS future for another week.
* BPS-FUT condition: Participants will practice BPS Future for two weeks.
* CONTROL condition: Participants will practice DAILY ACTIVITIES for two weeks.

DETAILED DESCRIPTION:
The design will permit two comparisons:

After the first week of the intervention, participants will answer the assessment. It will permit to compare BPS PAST, BPS FUTURE and CONTROL conditions (pre-post).

After the second week, participants will answer the assessment and then it will be possible to compare BPS PAST + BPS FUTURE combination, BPS FUTURE, and CONTROL conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years old or older.
* Participants must be willing to participate in the study.
* Participants must have a smartphone (Android or Ios).

Exclusion Criteria:

* To suffer from moderate depression or anxiety (scores of 11 or higher) measured by the Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983).
* To have "Flourishing mental health" measured by the Mental Health Continuum Short Form (MHC-SF; Keyes, 2009)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
Change of Positive and Negative Affect from baseline to post-intervention | Change from pre-intervention to post-intervention (2 weeks)
  Positive and Negative Affect Scale (PANAS; Watson, Clark & Tellegen, 1988)

SECONDARY OUTCOMES:
Wellbeing | Change from pre-intervention to post-intervention (2 weeks)
  The Mental Health Continuum Short Form (MHC-SF; Keyes, 2009)
Optimism | Change from pre-intervention to post-intervention (2 weeks)
  Life Orientation Test (LOT-R; Scheier, Carver & Bridges, 1994).
Satisfaction with life | Change from pre-intervention to post-intervention (2 weeks)
  Temporal Satisfaction with Life Scale (TSWLS; Pavot, Diener & Suh, 1998).
Self-efficacy | Change from pre-intervention to post-intervention (2 weeks)
  New General Self-efficacy Scale (NGSES; Chen, Gully & Eden, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Baños, PhD, Principal Investigator — University of Valencia
Locations (2):
- University of Twente, Enschede, Overijssel, Netherlands
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] King L. The Health Benefits of Writing About Life Goals. Personality and Social Psychology Bulletin 27(7): 798-807, 2001.
- [Background] Sheldon KM, Lyubomirsky S. How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology 1(2): 73-82, 2006.
- [Background] Peters ML, Flink IK, Boersma K, Linton SJ. Manipulating optimism: Can imagining a best possible self be used to increase positive future expectancies? The Journal of Positive Psychology 5(3): 204-211, 2010.